CLINICAL TRIAL: NCT02207777
Title: Weight Loss-Independent Metabolic Effects of Roux-En-Y Gastric Bypass in Diabetes
Acronym: RBD-T2D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 201403065; 1R01DK101578 (NIH)
Record Dates: First submitted 2014-07-31; First posted 2014-08-04 (Estimated); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Obesity; Type 2 Diabetes
Keywords: Obesity; Roux-en-Y gastric bypass (RYGB); Type 2 Diabetes; Weight Loss; Low-Calorie Diet
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2; Weight Loss | interventions — Caloric Restriction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Roux-en-Y gastric bypass (RYGB) (Experimental): Subjects in this group are scheduled to undergo roux-en-Y gastric bypass surgery to obtain approximately 16-18% (with a range of 16-25%) weight loss.
  Interventions: Procedure: Roux-en-Y gastric bypass surgery
- Low-calorie diet (Active Comparator): Subjects in this group will participate in a low-calorie diet intervention to obtain approximately 16-18% (with a range of 16-25%) weight loss.
  Interventions: Behavioral: Low-calorie diet

INTERVENTIONS:
Procedure: Roux-en-Y gastric bypass surgery — A surgical procedure to help subjects lose approximately 16-18% (with a range of 16-25%) of their body weight.
  Arms: Roux-en-Y gastric bypass (RYGB)
Behavioral: Low-calorie diet — Subjects will meet with a dietitian and/or behaviorist over approximately 6 months to lose approximately 16-18% (with a range of 16-25%) of their body weight.
  Arms: Low-calorie diet

SUMMARY:
For this purpose, we will compare the effects of targeted 16-18% (with a range of 16-25%) weight loss induced by Roux-en-Y Gastric bypass (RYGB) surgery with the same weight loss induced by a low-calorie diet (LCD) on liver and skeletal muscle insulin sensitivity, beta-cell function, and 24-hour metabolic homeostasis in obese subjects with or without T2D.

ELIGIBILITY:
Inclusion Criteria:

For RYGB group:

* Scheduled for this bariatric surgery
* Body Mass Index (BMI) 34-55 kg/m²
* Type 2 Diabetes
* Signed informed consent

For Low-Calorie Diet group:

* BMI 34-55 kg/m²
* Type 2 Diabetes and Non-Diabetics
* Signed informed consent

Exclusion Criteria:

For both RYGB & Low-Calorie Diet groups

* Regular use of tobacco products
* Previous intestinal resection
* Pregnant or breastfeeding
* Evidence of significant organ system dysfunction or disease other than T2D
* Use of any medication that might, in the opinion of the investigator, affect metabolic function
* Exercise ≥90 minutes per week

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Changes in hepatic insulin sensitivity | 6 months (before and after targeted weight loss)
  The outcome will be assessed by hyperinsulinemic-euglycemic-pancreatic-clamp procedure before and after weight loss.

SECONDARY OUTCOMES:
Changes in skeletal muscle and adipose tissue insulin sensitivity | 6 months (before and after targeted weight loss)
  The outcome will be assessed by hyperinsulinemic-euglycemic-pancreatic-clamp procedure before and after weight loss.
Changes in Beta-cell function | 6 months (before and after targeted weight loss)
  The outcome will be assessed as the product of beta-cell glucose sensitivity (ratio of post-meal insulin secretion rate to post-meal plasma glucose) during mixed-meal test and whole-body insulin sensitivity before and after weight loss.
Changes in glucose kinetics (glucose concentration and rate of appearance into the systemic circulation) in response to mixed-meal ingestion | 6 months (before and after targeted weight loss)
  The outcome will be measured by using dual glucose tracer mixed meal metabolic test and serial blood sampling for 4 hours before and after weight loss
Changes in 24-hour plasma glucose profile | 6 months (before and after targeted weight loss)
  The outcome will be determined by obtaining serial plasma glucose concentration measurements for 24 hours before and after weight loss
Changes in 24-hour plasma insulin profile | 6 months (before and after targeted weight loss)
  The outcome will determined by obtaining serial plasma insulin concentration measurements for 24 hours before and after weight loss
Changes in 24-hour plasma free fatty acid profile | 6 months (before and after targeted weight loss)
  The outcome will determined by obtaining serial plasma free fatty acid concentration measurements for 24 hours before and after weight loss
Changes in body fat mass | 6 months (before and after targeted weight loss)
  The outcome will be measured by using dual-energy X-ray absorptiometry before and after weight loss
Changes in intra-abdominal adipose tissue volume | 6 months (before and after targeted weight loss)
  The outcome will be measured by using magnetic resonance imaging before and after weight loss
Changes in intrahepatic triglyceride content | 6 months (before and after targeted weight loss)
  The outcome will be measured by using magnetic resonance imaging before and after weight loss
Changes in fat free mass | 6 months (before and after targeted weight loss)
  The outcome will be measured by using dual-energy X-ray absorptiometry before and after weight loss

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Klein, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Petersen MC, Yoshino M, Smith GI, Gaspar RC, Kahn M, Samovski D, Shulman GI, Klein S. Effect of Weight Loss on Skeletal Muscle Bioactive Lipids in People With Obesity and Type 2 Diabetes. Diabetes. 2024 Dec 1;73(12):2055-2064. doi: 10.2337/db24-0083. PMID 39264820
- [Background] Samovski D, Smith GI, Palacios H, Pietka T, Fuchs A, Patti GJ, Nawaz A, Kahn CR, Klein S. Effect of Marked Weight Loss on Adipose Tissue Biology in People With Obesity and Type 2 Diabetes. Diabetes Care. 2025 Aug 1;48(8):1342-1351. doi: 10.2337/dc24-2739. PMID 40208704
- [Background] Smith GI, Klein S. Plasma endotrophin levels correlate with insulin resistance in people with obesity. J Clin Invest. 2025 Apr 22;135(12):e190577. doi: 10.1172/JCI190577. eCollection 2025 Jun 16. No abstract available. PMID 40261704
- [Background] Yoshino M, Kayser BD, Yoshino J, Stein RI, Reeds D, Eagon JC, Eckhouse SR, Watrous JD, Jain M, Knight R, Schechtman K, Patterson BW, Klein S. Effects of Diet versus Gastric Bypass on Metabolic Function in Diabetes. N Engl J Med. 2020 Aug 20;383(8):721-732. doi: 10.1056/NEJMoa2003697. PMID 32813948
- [Derived] van Vliet S, Koh HE, Patterson BW, Yoshino M, LaForest R, Gropler RJ, Klein S, Mittendorfer B. Obesity Is Associated With Increased Basal and Postprandial beta-Cell Insulin Secretion Even in the Absence of Insulin Resistance. Diabetes. 2020 Oct;69(10):2112-2119. doi: 10.2337/db20-0377. Epub 2020 Jul 10. PMID 32651241